CLINICAL TRIAL: NCT01670253
Title: Randomized, Double-blind, Controlled, Parallel-group Study Reduction of Starvation Time Prior to Gastroscopy
Brief Title: Reduction of Starvation Time Prior to Gastroscopy
Acronym: RETIME
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough facilities to study
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Anton Bilenko, MD, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: S-20120069
Record Dates: First submitted 2012-08-14; First posted 2012-08-22 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Habile Adult Patients Referred to the Elective Gastroscopy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 2 (No Intervention): 6 hours of total fast for all solid and liquid food / drinks
- Group 1 (Experimental): * 6 hour fast from all solid foods and milk beverages
  * 2-hour thirst period before examination (patient may be in the period from 6 to 2 hours before the study drink any kind of clear liquids, ie liquids containing no milk products)
  * Approximately 2 hours before the time of examination please drink a glass (about 2 cups) clear sugary liquid - eg lemonade, apple juice, iced tea, soda or the like.
  Interventions: Behavioral: Group 1

INTERVENTIONS:
Behavioral: Group 1 — * 6 hour fast from all solid foods and milk beverages
  * 2-hour thirst period before examination (patient may be in the period from 6 to 2 hours before the study drink any kind of clear liquids, ie liquids containing no milk products)
  * Approximately 2 hours before the time of examination please drink a glass (about 2 cups) clear sugary liquid - eg lemonade, apple juice, iced tea, soda or the like.
  Arms: Group 1

SUMMARY:
The primary objective is to investigate whether intake of approximately 200 ml of sugary fluid 2 hours before the scheduled gastroscopy of the abdomen can reduce the discomfort of fasting period for patients without reducing the quality of the study.

Current standard for fasting and fluid intake before gastroscopy is completely fasting 6 hours before the study. Studies in patients in general anesthesia has been found that it does not increase the risk of aspiration of stomach content during the operation by allowing the patient to drink up to 2 hours prior to anesthesia induction. There are no studies that have examined the quality gastroscopy using this fasting procedure. Some studies show that intake of sugary liquids do not have significant effect on gastric emptying.

There are not deemed to be ethical problems with this study, as it seeks to show that a more lenient standard procedure in endoscopy is as safe as the established. The study is considered safe.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Sufficient knowledge of Danish to understand the written information
* legally competent patients

Exclusion Criteria:

* Patients with a history of pyloric stenosis (narrowing of the transition from stomach to the duodenum)
* Incapacitated patients
* Patients with daily vomiting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2014-12-11 (Actual)

PRIMARY OUTCOMES:
Number of uncomplicated examinations | participants will be followed for the duration of hospital stay, an expected average of 1 hour

SECONDARY OUTCOMES:
Reduction of discomfort for the patients according to the survey. | participants will be followed for the duration of hospital stay, an expected average of 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Anton Bilenko, MD, Principal Investigator — Odense University Hospital